CLINICAL TRIAL: NCT02562716
Title: A Randomized Phase II Study of Perioperative mFOLFIRINOX Versus Gemcitabine/Nab-Paclitaxel as Therapy for Resectable Pancreatic Adenocarcinoma
Brief Title: S1505: Combination Chemotherapy or Gemcitabine Hydrochloride and Paclitaxel Albumin-Stabilized Nanoparticle Formulation Before Surgery in Treating Patients With Pancreatic Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1505; NCI-2015-01236 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1505 (Other: SWOG); S1505 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Results first posted 2021-07-23 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Adenocarcinoma; Resectable Pancreatic Carcinoma
MeSH Terms: interventions — Fluorouracil; dehydroftorafur; Gemcitabine; Irinotecan; Oxaliplatin; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Pancreatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (mFOLFIRINOX, surgery) (Experimental): Patients receive oxaliplatin IV over 2 hours and irinotecan hydrochloride IV over 90 minutes on days 1 and 15. Patients also receive 5-fluorouracil IV over 46 hours on days 1-3 and 15-17. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of oxaliplatin, irinotecan hydrochloride, and fluorouracil treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Oxaliplatin; Procedure: Pancreatectomy
- Arm II (gemcitabine, nab-paclitaxel, and surgery) (Experimental): Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine hydrochloride treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation; Procedure: Pancreatectomy

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
  Arms: Arm I (mFOLFIRINOX, surgery)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
  Arms: Arm II (gemcitabine, nab-paclitaxel, and surgery)
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E
  Arms: Arm I (mFOLFIRINOX, surgery)
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
  Arms: Arm I (mFOLFIRINOX, surgery)
Drug: Paclitaxel Albumin-Stabilized Nanoparticle Formulation — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; nab-paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; protein-bound paclitaxel
  Arms: Arm II (gemcitabine, nab-paclitaxel, and surgery)
Procedure: Pancreatectomy — Undergo pancreatectomy
  Other Names: Excision of the Pancreas; Pancreas Excision

SUMMARY:
This randomized phase II trial studies how well fluorouracil, irinotecan hydrochloride, and oxaliplatin (combination chemotherapy) works and compares to gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation before surgery in treating patients with pancreatic cancer that can be removed by surgery. Drugs used in chemotherapy, such as fluorouracil, irinotecan hydrochloride, oxaliplatin, gemcitabine hydrochloride, and paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether combination chemotherapy is more effective than gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation before surgery in treating pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess 2-year overall survival in each treatment arm (fluorouracil, irinotecan hydrochloride, and oxaliplatin [modified (m)FOLFIRINOX] and gemcitabine [gemcitabine hydrochloride]/nab-paclitaxel [paclitaxel albumin-stabilized nanoparticle formulation]) in patients with resectable pancreatic cancer.

II. If the stated threshold is met in one or both arms: to choose the better regimen with respect to 2-year overall survival.

SECONDARY OBJECTIVES:

I. To estimate, for all patients and within treatment arms: frequency and severity of adverse events associated with chemotherapy in the perioperative setting.

II. To estimate, for all patients and within treatment arms: proportion of patients going to surgery for resection after preoperative chemotherapy.

III. To estimate, for all patients and within treatment arms: proportion of patients achieving macroscopically complete tumor removal with negative microscopic surgical margins (R0) resection after preoperative chemotherapy.

IV. To estimate, for all patients and within treatment arms: overall response rate following preoperative chemotherapy, including confirmed and unconfirmed, complete and partial response, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

V. To estimate, for all patients and within treatment arms: pathologic response rates after R0 or macroscopically complete tumor removal with any positive microscopic surgical margin (R1) resection.

VI. To estimate, for all patients and within treatment arms: patterns of recurrence (loco-regional, distant) after R0 or R1 resection.

VII. To estimate, for all patients and within treatment arms: disease-free survival from the time of R0 or R1 resection.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oxaliplatin intravenously (IV) over 2 hours and irinotecan hydrochloride IV over 90 minutes on days 1 and 15. Patients also receive fluorouracil IV over 46 hours on days 1-3 and 15-17. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of oxaliplatin, irinotecan hydrochloride, and fluorouracil treatment in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine hydrochloride treatment in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven pancreatic adenocarcinoma; histologies other than adenocarcinoma, or any mixed histologies, will NOT be eligible
* Patients must have measurable disease in the pancreas; computed tomography (CT) scans or magnetic resonance imaging (MRIs) used to assess measurable disease must have been completed within 28 days prior to registration; all disease must be assessed and documented on the baseline tumor assessment form
* Patients must have resectable primary tumor based on contrast-enhanced CT or MRI (CT or MRI without contrast as part of positron emission tomography [PET]/CT or PET/MRI is NOT acceptable; CT or MRI with contrast as part of PET/CT or PET/MRI is acceptable) of the chest, abdomen, and pelvis, where resectable is defined as:

  * No involvement of the celiac artery, common hepatic artery, and superior mesenteric artery (and, if present, replaced right hepatic artery)
  * No involvement, or < 180° interface between tumor and vessel wall, of the portal vein and/or superior mesenteric vein; and patent portal vein/splenic vein confluence
  * No evidence of metastatic disease
  * Note: for tumors of the body and tail of the pancreas, involvement of the splenic artery and vein of any degree is considered resectable disease
* CT scans or MRIs used to assess disease at baseline must be submitted for central review
* Patients must have surgical consult to verify patient is a surgical candidate within 21 days prior to registration
* Patients must not have received prior surgery, radiation therapy, chemotherapy, targeted therapy, or any investigational therapy for pancreatic cancer
* Patients must have a Zubrod performance status of 0-1
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x IULN
* Serum albumin >= 3 g/dL
* Serum creatinine =< IULN within 14 days prior to registration
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements will NOT be eligible
* No prior malignancy is allowed except for adequately treated basal (or squamous cell) skin cancer, in situ cervical cancer, in situ breast (ductal or lobular) cancer, or other cancer for which the patient has been disease and treatment-free for two years
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method for up to 3 months after the final administered dose of chemotherapy; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures, he/she is responsible for beginning contraceptive measures
* Sites must seek additional patient consent for the future use of specimens
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davendra Sohal, Principal Investigator — SWOG Cancer Research Network
Locations (807):
- United States (807):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arizona Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - University of California San Diego, San Diego, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Regional Cancer Center-Lee Memorial Health System, Fort Myers, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - The Watson Clinic, Lakeland, Florida
  - Jackson Memorial Hospital-Holtz Children's Hospital, Miami, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Baptist Health Corbin, Corbin, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Hardin Memorial Hospital, Elizabethtown, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Baptist Health Madisonville/Merle Mahr Cancer Center, Madisonville, Kentucky
  - Baptist Health Paducah, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Medical Center of Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - University Health-Conway, Monroe, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Frederick Memorial Hospital, Frederick, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Point, Grosse Pointe, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon and Rectal Association, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Hematology Oncology Consultants PC, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Hattiesburg Clinic - Hematology/Oncology Clinic, Hattiesburg, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Hematology Oncology Associates of Central New York-Onondaga Hill, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Cape Fear Cancer Specialists-Leland, Leland, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Cape Fear Cancer Specialists, Wilmington, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Salem Hospital, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Integrity Oncology PLLC-Collierville, Collierville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Ascension Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Sohal DPS, Boutin RD, Lenchik L, Kim J, Beg MS, Wang-Gillam A, Wade JL 3rd, Guthrie KA, Chiorean EG, Ahmad SA, Lowy AM, Philip PA, Chang VT. Body composition measurements and clinical outcomes in patients with resectable pancreatic adenocarcinoma - analysis from SWOG S1505. J Gastrointest Surg. 2024 Mar;28(3):232-235. doi: 10.1016/j.gassur.2023.12.022. Epub 2024 Jan 19. PMID 38445914
- [Derived] Sohal DPS, Duong M, Ahmad SA, Gandhi NS, Beg MS, Wang-Gillam A, Wade JL 3rd, Chiorean EG, Guthrie KA, Lowy AM, Philip PA, Hochster HS. Efficacy of Perioperative Chemotherapy for Resectable Pancreatic Adenocarcinoma: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 Mar 1;7(3):421-427. doi: 10.1001/jamaoncol.2020.7328. PMID 33475684
- [Derived] Ahmad SA, Duong M, Sohal DPS, Gandhi NS, Beg MS, Wang-Gillam A, Wade JL 3rd, Chiorean EG, Guthrie KA, Lowy AM, Philip PA, Hochster HS. Surgical Outcome Results From SWOG S1505: A Randomized Clinical Trial of mFOLFIRINOX Versus Gemcitabine/Nab-paclitaxel for Perioperative Treatment of Resectable Pancreatic Ductal Adenocarcinoma. Ann Surg. 2020 Sep 1;272(3):481-486. doi: 10.1097/SLA.0000000000004155. PMID 32740235

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 147 participants were randomized, but 43 were found to be ineligible per central radiology review, and 1 was found to be ineligible due to incorrect primary tumor. One patient withdrew study consent prior to any therapy and was not evaluable. Therefore 102 were deemed eligible and analyzable for the primary analysis.
Groups:
- mFOLFIRINOX ->Surg ->mFOLFIRINOX: Patients receive oxaliplatin IV over 2 hours and irinotecan hydrochloride IV over 90 minutes on days 1 and 15. Patients also receive 5-fluorouracil IV over 46 hours on days 1-3 and 15-17. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of oxaliplatin, irinotecan hydrochloride, and fluorouracil treatment in the absence of disease progression or unacceptable toxicity.
- Gem/Nab-P ->Surg ->Gem/Nab-P: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine hydrochloride treatment in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | mFOLFIRINOX ->Surg ->mFOLFIRINOX | Gem/Nab-P ->Surg ->Gem/Nab-P
Started | 55 | 47
Participants Assessed for AEs | 53 | 45
Completed | 27 | 19
Not Completed | 28 | 28
Not completed — Adverse Event | 7 | 14
Not completed — Withdrawal unrelated to AE | 7 | 1
Not completed — Progression | 8 | 10
Not completed — Death | 2 | 1
Not completed — Not protocol specified | 4 | 2

BASELINE CHARACTERISTICS:
Population: 147 participants were randomized, but 43 were found to be ineligible per central radiology review, and 1 was found to be ineligible due to incorrect primary tumor. One patient withdrew study consent prior to any therapy and was not evaluable. Therefore 102 were deemed eligible and analyzable for the primary analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | mFOLFIRINOX ->Surg ->mFOLFIRINOX | Gem/Nab-P ->Surg ->Gem/Nab-P | Total
Number analyzed (Participants) | 55 | 47 | 102
Age, Continuous [Median (Full Range); unit: years] | 66 [44 to 76] | 64 [46 to 75] | 64 [44 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 36 | 24 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 51 | 43 | 94
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 52 | 39 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Zubrod Performance Status [Count of Participants; unit: Participants] — Scale: 0-5, with 0 denoting perfect health and 5 death.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    0 | 34 | 31 | 65
    1 | 21 | 16 | 37

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is the length of time between protocol registration and patient death
Time Frame: Up to 4 years for the estimates of median overall survival. Up to 2 years for Statistical Analysis 1 and 2, comparing the observed 2-year overall survival (OS) to the null hypothesis of 40%, in each arm.
Population: Eligible and analyzable participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mFOLFIRINOX ->Surg ->mFOLFIRINOX | Gem/Nab-P ->Surg ->Gem/Nab-P
Number analyzed (Participants) | 55 | 47
Months | 23.2 [17.6 to 45.9] | 23.6 [17.8 to 31.7]
Statistical Analysis 1: Comparison: mFOLFIRINOX ->Surg ->mFOLFIRINOX; For each arm, the observed 2-year overall survival (OS) was compared to the null hypothesis of 40%, assuming a 58% alternative hypothesis, 88% power, and a 1-sided significance of 0.05; Test type: Superiority; p = .15, Log Rank
Statistical Analysis 2: Comparison: Gem/Nab-P ->Surg ->Gem/Nab-P; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .14, Log Rank

2. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Only adverse events that are possibly, probably or definitely related to preoperative and postoperative chemotherapy are reported.
Time Frame: Duration of treatment and follow up until death or 4 years post registration.
Population: Participants who received at least one dose of protocol treatment and were thus eligible for AE assessment.
Measure: Number; unit: Participants
Groups:
- mFOLFIRINOX->Surg->mFOLFIRINOX: Patients receive oxaliplatin IV over 2 hours and irinotecan hydrochloride IV over 90 minutes on days 1 and 15. Patients also receive 5-fluorouracil IV over 46 hours on days 1-3 and 15-17. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of oxaliplatin, irinotecan hydrochloride, and fluorouracil treatment in the absence of disease progression or unacceptable toxicity.
- Gem/Nab-P->Surg->Gem/Nab-P: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine hydrochloride treatment in the absence of disease progression or unacceptable toxicity.
Arm/Group | mFOLFIRINOX->Surg->mFOLFIRINOX | Gem/Nab-P->Surg->Gem/Nab-P
Number analyzed (Participants) | 53 | 45
Participants
  Abdominal infection | 1 | 0
  Acute kidney injury | 0 | 1
  Alanine aminotransferase increased | 3 | 2
  Allergic reaction | 1 | 0
  Anemia | 4 | 4
  Anorexia | 2 | 0
  Aspartate aminotransferase increased | 2 | 1
  Biliary tract infection | 0 | 1
  Blood bilirubin increased | 1 | 3
  Colonic perforation | 0 | 1
  Constipation | 0 | 1
  Dehydration | 1 | 0
  Diarrhea | 8 | 3
  Dysesthesia | 1 | 0
  Dyspnea | 0 | 1
  Fall | 1 | 0
  Fatigue | 4 | 3
  Febrile neutropenia | 0 | 2
  Hepatobiliary disorders - Other, specify | 1 | 0
  Hyperglycemia | 2 | 2
  Hypertension | 0 | 1
  Hypoalbuminemia | 0 | 1
  Hypoglycemia | 0 | 1
  Hypokalemia | 3 | 1
  Hypomagnesemia | 0 | 2
  Hyponatremia | 2 | 2
  Infections and infestations - Other, specify | 1 | 1
  Infusion related reaction | 1 | 0
  Insomnia | 0 | 1
  Leukocytosis | 1 | 0
  Lung infection | 1 | 2
  Lymphocyte count decreased | 0 | 2
  Mucositis oral | 0 | 1
  Myocardial infarction | 1 | 0
  Nausea | 3 | 1
  Neutrophil count decreased | 11 | 17
  Non-cardiac chest pain | 0 | 1
  Pancreatitis | 1 | 0
  Papulopustular rash | 0 | 1
  Peripheral motor neuropathy | 1 | 0
  Peripheral sensory neuropathy | 5 | 3
  Platelet count decreased | 3 | 2
  Pneumonitis | 0 | 1
  Rectal hemorrhage | 0 | 1
  Respiratory failure | 0 | 1
  Sepsis | 1 | 2
  Skin infection | 1 | 0
  Thromboembolic event | 2 | 0
  Vomiting | 2 | 0
  Weight loss | 2 | 0
  White blood cell decreased | 1 | 6

3. Secondary Outcome: Number of Patients Going to Surgery for Resection After Preoperative Chemotherapy.
Time Frame: Up to 8 months post registration (and within 4 to 8 weeks after the last dose of Cycle 3 preoperative chemotherapy).
Population: Eligible and analyzable participants
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFIRINOX ->Surg ->mFOLFIRINOX | Gem/Nab-P ->Surg ->Gem/Nab-P
Number analyzed (Participants) | 55 | 47
Participants | 40 | 33

4. Secondary Outcome: Number of Patients Achieving R0 Resection After Preoperative Chemotherapy.
Description: R0 resection classification is defined as macroscopically complete tumor removal with negative microscopic surgical margins (bile duct, pancreatic parenchyma, and superior mesenteric artery margins).
Time Frame: Up to 8 months post registration (and within 4 to 8 weeks after the last dose of Cycle 3 preoperative chemotherapy).
Population: Eligible and analyzable participants undergoing surgical resection.
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFIRINOX ->Surg ->mFOLFIRINOX | Gem/Nab-P ->Surg ->Gem/Nab-P
Number analyzed (Participants) | 40 | 33
Participants | 34 | 28

5. Secondary Outcome: Number of Participants With a Response Following Preoperative Chemotherapy, Including Confirmed and Unconfirmed, Complete and Partial Response, Per RECIST 1.1.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 6 months post registration (and within 2 to 4 weeks after the last dose of Cycle 3 preoperative chemotherapy.).
Population: Eligible and analyzable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFIRINOX ->Surg ->mFOLFIRINOX | Gem/Nab-P ->Surg ->Gem/Nab-P
Number analyzed (Participants) | 55 | 47
Participants | 5 | 10

6. Secondary Outcome: Number of Participants With Complete Response, Moderate Response, Minimal Response, and Poor or No Response After Resection.
Description: Pathologic response was evaluated after the patient had surgery, and was based on local pathology review of the resected surgical specimen, according to the following Tumor Regression Grade definitions:
  0: Complete response - no residual tumor
  1. Moderate response - minimal residual cancer (single cells or small groups of cancer cells)
  2. Minimal response - residual cancer outgrown by fibrosis
  3. Poor or no response - no definite response identified (minimal or no tumor kill; extensive residual cancer)
Time Frame: Up to 8 months post registration (and within 4 to 8 weeks after the last dose of Cycle 3 preoperative chemotherapy).
Population: Eligible and analyzable participants undergoing resection.
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFIRINOX ->Surg ->mFOLFIRINOX | Gem/Nab-P ->Surg ->Gem/Nab-P
Number analyzed (Participants) | 40 | 33
Participants
  Complete Response | 1 | 3
  Moderate Response | 9 | 10
  Minimal Response | 12 | 10
  Poor or No Response | 18 | 10

7. Secondary Outcome: Number of Participants With Loco-regional and Distant Recurrence After R0 or R1 Resection.
Description: Loco-regional recurrence is defined as any evidence of new disease within the pancreatic tumor bed based on surveillance scans. The pancreatic tumor bed includes:
  1. Superior mesenteric artery and vein lymph nodes
  2. Lymph nodes in porta hepatis (bile duct, portal vein, hepatic artery lymph nodes)
  3. Lymph nodes around left renal vein, inferior vena cava or aorta
  4. Celiac axis lymph nodes.
  Distant Recurrence is defined as any evidence of new disease outside the primary tumor bed (liver, lungs, etc.) based on surveillance scans.
Time Frame: Up to 4 years
Population: Eligible and analyzable participants undergoing resection.
Measure: Count of Participants; unit: Participants
Arm/Group | mFOLFIRINOX ->Surg ->mFOLFIRINOX | Gem/Nab-P ->Surg ->Gem/Nab-P
Number analyzed (Participants) | 40 | 33
Participants
  No Progression | 13 | 17
  Loco-regional recurrence | 9 | 4
  Distant recurrence | 13 | 9
  Both loco-regional and distant recurrence | 5 | 2
  Not assessed due to death (cardiac arrest) prior to start of post-op chemo | 0 | 1

8. Secondary Outcome: Disease-free Survival From the Time of R0 or R1 Resection.
Description: Disease-free survival (DFS) is calculated for patients who undergo surgical resection (R0/R1). DFS will be measured from the date of surgical resection to date of first documentation of recurrence (loco-regional or distant) or death due to any cause. Patients last known to be alive and free of disease will be censored at date of last contact.
Time Frame: Up to 4 years
Population: Eligible and analyzable participants undergoing surgical resection.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | mFOLFIRINOX ->Surg ->mFOLFIRINOX | Gem/Nab-P ->Surg ->Gem/Nab-P
Number analyzed (Participants) | 40 | 33
Months | 10.9 [8.7 to 16.6] | 14.2 [7.3 to 18.6]

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 4 years post registration.
Description: Adverse Events (AEs) are reported by CTCAE Version 5.0.
Groups:
- mFOLFIRINOX->Surg->mFOLFIRINOX: Patients receive oxaliplatin IV over 2 hours and irinotecan hydrochloride IV over 90 minutes on days 1 and 15. Patients also receive 5-fluorouracil IV over 46 hours on days 1-3 and 15-17. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of oxaliplatin, irinotecan hydrochloride, and fluorouracil treatment in the absence of disease progression or unacceptable toxicity.
  Participants who received at least one dose of protocol treatment and were thus eligible for AE assessment are included in the Serious Adverse Events and Other Adverse Events tables. All eligible participants were assessed for All-Cause Mortality.
- Gem/Nab-P->Surg->Gem/Nab-P: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable disease or better undergo pancreatectomy 4-8 weeks after completion of first 3 courses of treatment. Within 4-8 weeks following pancreatectomy, patients receive an additional 3 courses of paclitaxel albumin-stabilized nanoparticle formulation and gemcitabine hydrochloride treatment in the absence of disease progression or unacceptable toxicity.
  Participants who received at least one dose of protocol treatment and were thus eligible for AE assessment are included in the Serious Adverse Events and Other Adverse Events tables. All eligible participants were assessed for All-Cause Mortality.
Arm/Group | mFOLFIRINOX->Surg->mFOLFIRINOX | Gem/Nab-P->Surg->Gem/Nab-P
All-Cause Mortality (participants affected / at risk) | 32/55 | 32/47
Serious Adverse Events (participants affected / at risk) | 3/53 | 5/45
Other Adverse Events (participants affected / at risk) | 53/53 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFIRINOX->Surg->mFOLFIRINOX (N=53) | Gem/Nab-P->Surg->Gem/Nab-P (N=45)
Cardiac arrest (Cardiac disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Hepatobiliary disorders-Other (Hepatobiliary disorders) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFIRINOX->Surg->mFOLFIRINOX (N=53) | Gem/Nab-P->Surg->Gem/Nab-P (N=45)
Anemia (Blood and lymphatic system disorders) | 32 | 37
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 3 | 6
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0
Blurred vision (Eye disorders) | 4 | 0
Dry eye (Eye disorders) | 2 | 1
Eye disorders-Other (Eye disorders) | 3 | 4
Eye pain (Eye disorders) | 1 | 3
Watering eyes (Eye disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 24 | 22
Anal pain (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 3 | 6
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 15 | 16
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 39 | 29
Dry mouth (Gastrointestinal disorders) | 2 | 3
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 6 | 7
Dysphagia (Gastrointestinal disorders) | 3 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 4 | 3
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 4 | 5
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 2
Gastroparesis (Gastrointestinal disorders) | 2 | 3
Hemorrhoids (Gastrointestinal disorders) | 3 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Malabsorption (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 7 | 6
Nausea (Gastrointestinal disorders) | 38 | 29
Oral pain (Gastrointestinal disorders) | 1 | 1
Pancreatic fistula (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 17 | 16
Chills (General disorders) | 8 | 9
Edema limbs (General disorders) | 3 | 10
Fatigue (General disorders) | 41 | 38
Fever (General disorders) | 10 | 14
Flu like symptoms (General disorders) | 2 | 8
Gait disturbance (General disorders) | 1 | 0
General disorders and admin site conditions - Other (General disorders) | 1 | 2
Hypothermia (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 5 | 1
Irritability (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 2
Malaise (General disorders) | 3 | 4
Neck edema (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 3 | 1
Pain (General disorders) | 7 | 13
Bile duct stenosis (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Allergic reaction (Immune system disorders) | 4 | 0
Abdominal infection (Infections and infestations) | 1 | 1
Biliary tract infection (Infections and infestations) | 0 | 2
Bronchial infection (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Gum infection (Infections and infestations) | 0 | 1
Infections and infestations-Other (Infections and infestations) | 3 | 2
Lung infection (Infections and infestations) | 1 | 4
Mucosal infection (Infections and infestations) | 1 | 0
Papulopustular rash (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 4
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 5 | 4
Upper respiratory infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Wound infection (Infections and infestations) | 3 | 4
Biliary anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastric anastomotic leak (Injury, poisoning and procedural complications) | 0 | 1
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 23 | 17
Alkaline phosphatase increased (Investigations) | 25 | 16
Aspartate aminotransferase increased (Investigations) | 21 | 17
Blood bilirubin increased (Investigations) | 6 | 8
Cholesterol high (Investigations) | 1 | 0
Creatinine increased (Investigations) | 4 | 7
INR increased (Investigations) | 0 | 2
Investigations-Other (Investigations) | 4 | 3
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 6 | 7
Neutrophil count decreased (Investigations) | 25 | 31
Pancreatic enzymes decreased (Investigations) | 1 | 2
Platelet count decreased (Investigations) | 20 | 27
Weight gain (Investigations) | 3 | 1
Weight loss (Investigations) | 21 | 11
White blood cell decreased (Investigations) | 15 | 24
Anorexia (Metabolism and nutrition disorders) | 24 | 22
Dehydration (Metabolism and nutrition disorders) | 9 | 7
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 18 | 14
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 25 | 18
Hypocalcemia (Metabolism and nutrition disorders) | 11 | 11
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 21 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 10 | 5
Hyponatremia (Metabolism and nutrition disorders) | 11 | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 6
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 14
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Ataxia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 10 | 6
Dysarthria (Nervous system disorders) | 1 | 0
Dysesthesia (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 11 | 8
Dysphasia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 7 | 8
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Movements involuntary (Nervous system disorders) | 1 | 0
Nervous system disorders-Other (Nervous system disorders) | 5 | 1
Paresthesia (Nervous system disorders) | 6 | 0
Peripheral motor neuropathy (Nervous system disorders) | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 28 | 19
Sinus pain (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Spasticity (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 7 | 7
Confusion (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 6 | 11
Hallucinations (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 5 | 12
Restlessness (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 0
Renal calculi (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 1
Genital edema (Reproductive system and breast disorders) | 0 | 2
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 7
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 | 3
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 | 0
Flushing (Vascular disorders) | 1 | 1
Hot flashes (Vascular disorders) | 1 | 3
Hypertension (Vascular disorders) | 8 | 11
Hypotension (Vascular disorders) | 8 | 8
Superficial thrombophlebitis (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 6 | 3
Vascular disorders-Other (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/16/NCT02562716/Prot_SAP_ICF_000.pdf